CLINICAL TRIAL: NCT04064710
Title: The Biological Allograft Chain Tissue Implant & Associated Manual Surgical Instrumentation: A Prospective, Post-Market Study
Brief Title: Biological Allograft Chain Tissue Implant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lenoss Medical (Industry)
Collaborators: MCRA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP-18-001
Record Dates: First submitted 2019-08-20; First posted 2019-08-22 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Vertebral Body Compression Fracture(s)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Allograft Tissue (Other): Allograft tissue product for patients with painful vertebral compression fractures
  Interventions: Procedure: Vertebral Body Augmentation; Device: Manual Surgical Instruments

INTERVENTIONS:
Procedure: Vertebral Body Augmentation — Use allograft tissue in patients with one or two level, thoracic or lumbar T6-L5, vertebral compression fractures.
Device: Manual Surgical Instruments — Lenoss Medical manual surgical access and cavity creation instruments will be used when implanting the allograft tissue.

SUMMARY:
A prospective, multi-center study evaluating allograft tissue as a bone void filler when implanted with Lenoss Medical manual surgical instrumentation in patients with painful vertebral compression fractures.

DETAILED DESCRIPTION:
Vertebral compression fractures can be associated with instability and severe, persistent pain and limitation of activities. This post market study is being conducted to assess fracture stability over time.

ELIGIBILITY:
Inclusion Criteria:

1. Skeletally mature adult ≥ 50 years of age at the time of surgery;
2. Currently in an independent living environment;
3. One- or two- level, acute (within six weeks of injury), thoracic or lumbar (T6-L5) vertebral body compression fracture(s) with evidence of marrow edema by MRI/CT;
4. Adequate vertebral body height and geometry for insertion of the access instruments, as determined by the investigator and suitable candidate for standard kyphoplasty or vertebroplasty procedure;
5. VAS back pain score ≥ 70 mm on a 100 mm scale;
6. Has central pain over the spinous process upon palpation at the planned vertebral index level;
7. Has failed prior non-surgical medical management (i.e. - physical therapy, narcotic and/or non-narcotic medication)
8. Psychosocially, mentally and physically able to fully comply with this protocol including adhering to scheduled visits, treatment plan, completing forms, and other study procedures;
9. Personally signed and dated informed consent document prior to any study-related procedures indicating that the patient has been informed of all pertinent aspects of the study.

Exclusion Criteria:

1. More than two levels with a vertebral compression fracture;
2. Previous treated or untreated vertebral compression fracture at the to be treated level(s);
3. Uncorrectable coagulopathy;
4. Previous instrumented spinal surgery;
5. Significant vertebral collapse defined as > 70% of original vertebral height, or a burst, or pedicle fracture;
6. Degenerative scoliosis, defined as Cobb angle > 20° at any level;
7. Pre-existing neurological deficit or radicular pain that is not well defined or unstable;
8. Disabling back pain secondary to causes other than acute fracture;
9. Inability to walk or stand prior to sustaining the vertebral compression fracture;
10. Active systemic or local infection;
11. Known history of Paget's disease, osteomalacia, or any other metabolic bone disease;
12. Morbid obesity defined as a body mass index > 40 kg/m2;
13. Active malignancy. A patient with a history of any invasive malignancy (except nonmelanoma skin cancer), unless treated with curative intent and there has been no clinical signs or symptoms of the malignancy for more than 5 years;
14. Current or recent history (within last 2 years) of substance abuse (e.g., recreational drugs, narcotics, or alcohol);
15. Currently involved in study of another investigational product that may affect outcome;
16. History of psychosocial disorders that could prevent accurate completion of self reporting assessment scales;
17. Pregnant or planning to become pregnant during the study period;
18. Involved in active spinal litigation;
19. Involved in a workers compensation case;
20. Prisoner or ward of the state;
21. Unable to undergo a MRI/CT procedure.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2019-06-10 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate fracture stability assessed via subject- reported pain over time | 12 months
  Subject-reported pain over time using the allograft tissue will be assessed using the Visual Analog Scale (VAS) for back pain on a scale of 0mm (no pain) to 100mm (worst pain imaginable).

SECONDARY OUTCOMES:
Measure of Physical Disability Assessed via the Roland Morris Disability Questionnaire | 12 months
  The Roland Morris Disability Questionnaire is a widely used health status measure for physical disability caused by low back pain. Scores range from 0 to 24 with higher scores representing higher levels of pain-related disability.
Measurement of Quality of Life Assessed via the EuroQol Health Outcome Instrument (EQ-5D-3L) | 12 months
  The EQ-5D-3L is a standardized instrument used as a measure of health outcomes. It contains questions in 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and provides a simple descriptive profile and single index for health status preference. In addition, there is a Visual Analog Scale (VAS). The VAS is the participant's rating of their health on a scale of 0 "worst imaginable health state" to 100 "best imaginable health state".
Measurement of Activities of Daily Living Assessed via the Modified Tegner Activity Level Scale | 12 months
  The Modified Tegner Activity Level Scale is designed to measure a patient's activities of daily living, recreation, and competitive sports. The scale includes an assessment of level of activity pre- and post- injury. The scores range from 0 to 10 with a 0 representing sick leave or disability.
Frequency of Implant Related Complications | 12 months
  The frequency of allograft tissue related complications will be tabulated. Intra-operative complications, surgical time, and any other significant adverse events will be summarized as safety variables. Adverse events will be tabulated by physician's assessment of seriousness, severity, expectedness, the event's causative relation to the allograft tissue or the Access and Cavity Creation instruments, and by elapsed time since surgery. Adverse events that require secondary surgical intervention (SSI) will be flagged.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Colorado Denver | Anschutz Medical Campus, Denver, Colorado
  - North Shore University Hospital, Manhasset, New York
  - Mount Sinai, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Clinical Investigations LLC, Edmond, Oklahoma

IPD SHARING:
Plan to Share IPD: No